CLINICAL TRIAL: NCT02022423
Title: Physical Activity Daily - An Internet-Based Walking Program for Patients With Peripheral Arterial Disease
Acronym: PAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Elizabeth Anne Jackson, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NCT02022423
Record Dates: First submitted 2013-12-05; First posted 2013-12-27 (Estimated); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Peripheral Arterial Disease
Keywords: peripheral arterial disease; walking; eHealth; telehealth
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: Four groups are included in this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Telephone Counseling (Active Comparator): Weekly telephone calls to assess compliance to exercise prescription and discuss various topics related to adoption and adherence to walking programs
  Interventions: Behavioral: Telephone counseling
- Internet-based walking program (Experimental): Weekly automated goals are delivered via email to subject; goals are based on previous week's step count accumulation.
  Interventions: Behavioral: Internet-based walking program
- Telephone counseling and Internet-based walking program (Experimental): Weekly telephone calls to assess compliance to exercise prescription and discuss various topics related to adoption and adherence to walking programs plus weekly automated goals are delivered via email to subject; goals are based on previous week's step count accumulation.
  Interventions: Behavioral: Telephone counseling; Behavioral: Internet-based walking program
- Usual Care (No Intervention): Subjects will continue with their health care as usual

INTERVENTIONS:
Behavioral: Telephone counseling — 4 months of weekly contact to update exercise prescription and discuss barriers and challenges to adherence
  Arms: Telephone Counseling; Telephone counseling and Internet-based walking program
Behavioral: Internet-based walking program — Four-month Internet-based walking program consisting of weekly step count goals
  Arms: Internet-based walking program; Telephone counseling and Internet-based walking program

SUMMARY:
Peripheral arterial disease (PAD) is a significant vascular condition affecting millions of adults. Exercise such as walking is highly effective for reducing PAD symptoms such as claudication (pain with walking) and improving physical function. The trial examines the efficacy of a internet-delivered walking program for patients with PAD. Comparator groups including telephone counselling, the combination of internet-delivered walking program + telephone counseling, or usual care. The primary outcome of interest is maximal walking distance.

DETAILED DESCRIPTION:
With the aging of the American population, the numbers of adults with peripheral arterial disease (PAD) will increase significantly over the next several decades. Patients with PAD are at increased risk for morbidity and mortality including both cardiovascular and all-cause mortality. While regular physical activity reduces risk for vascular events and is recommended for treatment of PAD patients, few patients meet recommended goals. Exercise programs which increase long-term adherence to walking can be an important contribution to PAD treatment. Our Internet-based intervention, builds on a walking enhancement program developed by members of our team and is shown to improve adherence among patients with vascular disease such as coronary artery disease (CAD). Using a randomized, controlled trial study design, we propose to test an automated Internet-based walking program to improve long-term adherence to walking while increasing walking distance, and health-related quality of life, among patients with PAD. Participants will be randomized to 1 of four study groups: 1) weekly telephone counseling, 2) an Internet-based walking program, 3) a combination of telephone counseling and Internet-based walking program, or 4) a usual care group. The Internet-based walking program has been shown to increase both adherence to walking and overall walking duration in populations with chronic complex conditions such as CAD and diabetes. There is a strong need to develop interventions, easily generalizable to a real-world population, to improve the reach of lifestyle interventions which result in improved physical function and adherence to regular exercise among complex medical patients. Patients such as those with PAD (a CAD risk equivalent) stand to benefit the most from such programs.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 40

Diagnosis of PAD due to atherosclerosis, documented by 1 or more of the following:

* documented ankle brachial index (ABI) ≤ 0.9 in at least one leg
* toe brachial index ≤ .70 for participants with an ABI > 1.3
* documented arterial disease by MRI, CT or angiogram Ability to walk at least 150 feet without the assistance of a cane or walker. Are sedentary (defined as < 150 minutes per week of physical activity). Able to obtain medical clearance from a primary care provider, cardiologist, vascular specialist, endocrinologist, nurse practitioner, or physician assistant.

Competent to give informed consent. Have regular access to a computer with an Internet connection that allows software downloading.

Be a regular email user (check email at least once a week).

Exclusion Criteria:

PAD due to non-atherosclerotic causes such as trauma, entrapment syndromes or congenital anomalies.

No primary provider, or cardiologist or vascular provider Life expectancy of under 1-year Co-morbidities which limit physical activity to a severe degree (defined as the inability to walk a grocery store aisle unassisted) Signs of critical limb ischemia and/or planned peripheral revascularization in the next 12-months

A diagnoses of any of the following cardiovascular events in the past 3 months:

* stroke/transient ischemic attack
* myocardial infarction
* unstable angina
* percutaneous coronary intervention
* coronary bypass graft surgery A diagnoses of any of the following cardiovascular conditions
* severe valve disease untreated
* complex arrhythmia untreated
* New York Heart Association class III-IV heart failure Current substance abuse, or significant psychiatric disorder, or dementia which limits the participant's ability to follow the study protocol Pregnancy Non-English speaking

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Change in maximal walking distance | Baseline to 4 months
  measured using the Gardner-Skinner protocol treadmill test, noting time to moderate claudication
Change in PAD-specific health-related quality of life | Baseline to 4 months
  measured using disease specific Peripheral Artery Questionnaire (PAQ) which uses scale scores of 0 to 100, with high numbers indicating better outcomes.
Change in general health-related quality of life | Baseline to 4 months
  measured using the EuroQol 5 Dimension Scale (EQ-5D) which is comprised of a descriptive system questionnaire containing 5 questions and a visual analogue scale ranging from 0 to 100 with 0 being worse health state imaginable and 100 being best health state imaginable. The descriptive system questionnaire is scored by assigning a 1-digit number to the participant's answer choice for each of the 5 questions, then combining each into a 5-digit number indicating their health state.
Change in global health-related quality of life | Baseline to 4 months
  measured using the Patient Reported Outcomes Measurement Information System (PROMIS) Questionnaire that includes questions from physical, mental, and social health domains and is scored using a T-score metric. A higher score equals more of a concept being measured which can indicate better or worse outcomes depending on the concept being measured.

SECONDARY OUTCOMES:
Change in pain-free walking distance | Baseline to 4 months
  measured using the Gardner-Skinner protocol treadmill test, time to onset of claudication
Change in maximal walking distance | Baseline to 12 months
  measured using the Gardner-Skinner protocol treadmill test, noting time to moderate claudication
Change in PAD-specific health-related quality of life | Baseline to 12 months
  measured using disease specific Peripheral Artery Questionnaire (PAQ) which uses scale scores of 0 to 100, with high numbers indicating better outcomes.
Change in general health-related quality of life | Baseline to 12 months
  measured using EuroQol 5 Dimension Scale (EQ-5D) which is comprised of a descriptive system questionnaire containing 5 questions and a visual analogue scale ranging from 0 to 100 with 0 being worse health state imaginable and 100 being best health state imaginable. The descriptive system questionnaire is scored by assigning a 1-digit number to the participant's answer choice for each of the 5 questions, then combining each into a 5-digit number indicating their health state.
Change in global health-related quality of life | Baseline to 12 months
  measured using the Patient Reported Outcomes Measurement Information System (PROMIS) Questionnaire that includes questions from physical, mental, and social health domains and is scored using a T-score metric. A higher score equals more of a concept being measured which can indicate better or worse outcomes depending on the concept being measured.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A. Jackson, MD MPH FACC, Principal Investigator — University of Alabama at Birmingahm
Locations (2):
- United States (2):
  - University of Alabama Birmingham, Birmingham, Alabama
  - University of Michigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kumar AM, Lyden AK, Carlozzi NE, Sen A, Richardson CR, Jackson EA. The Physical Activity Daily (PAD) Trial: The rationale and design of a randomized controlled trial evaluating an internet walking program to improve maximal walking distance among patients with peripheral arterial disease. Contemp Clin Trials. 2018 Apr;67:23-30. doi: 10.1016/j.cct.2017.12.009. Epub 2017 Dec 21. PMID 29274894
- [Derived] Jones R, Enogela EM, Zumbro EL, Soukhamneut P, Richardson CR, Buford TW, Jackson EA. Assessment of Frailty Among Older Adults in the Physical Activity Daily Trial. J Appl Gerontol. 2024 Oct;43(10):1428-1437. doi: 10.1177/07334648241244690. Epub 2024 Apr 24. PMID 38655762